CLINICAL TRIAL: NCT05324878
Title: HIGHway Project: Honoring Individual Goals and Hopes: Implementing Advance Care Planning for Persons With Kidney Disease on Dialysis
Brief Title: Honoring Individual Goals and Hopes: Implementing Advance Care Planning for Persons With Kidney Disease on Dialysis
Acronym: HIGHway
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Medical Technology and Practice Patterns Institute (Unknown); Western Carolina University (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: NCR213481; DI-2020C2-20362 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2022-03-11; First posted 2022-04-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Kidney Diseases; Kidney Failure
Keywords: advance care planning; social workers; implementation research; patient-centered care; shared decision-making; nurses
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Population 1: Social workers/Nurses: Social workers and nurses working at participating dialysis centers. Dialysis centers will be selected based on demographic data of the center (urbanicity, population served, size of center, patients treated, etc) to provide for diversity of centers participating.
  Interventions: Other: Training
- Population 2a: Patients receiving care at the dialysis center: 2a. When an advance care planning conversation takes place, social worker/nurse will provide patient with an informational flyer about the HIGHway project and a postcard.
- Population 2b: Patients receiving care at the dialysis center: 2b. Social worker/nurse will identify one patient willing to have a recording made of advance care planning conversation between social worker/nurse and patient.

INTERVENTIONS:
Other: Training — Social workers/nurses participants are agreeing to participating in the training program (3 sessions of 2 hours over a period of six weeks - one session every 2 weeks), follow up training sessions (occurring monthly), mentorship calls with social worker faculty on the project team, recording one conversation between social worker and a patient for quality improvement purposes, and completing evaluation of the project interventions (5-minute questionnaire after each education session, 15-minute questionnaire at end of participation in project).
  Groups: Population 1: Social workers/Nurses

SUMMARY:
The PCORI HIGHway project name embodies its goal: the way to "Honor Individuals Goals and Hopes". HIGHway trains and supports dialysis center social workers and nurses to communicate with their patients about their hopes and goals for their future care plans. This process, known as advance care planning (ACP), helps relieve patient concerns about the future, lays the foundation for better goal-concordant care at the end of life, and fosters deeper connection between patient and the dialysis care team. The HIGHway project will provide training and ongoing coaching to social workers and other change team members at 50-60 dialysis centers throughout the US. The goal is to integrate advance care planning conversations between dialysis patients and their health care team into the ongoing workflow of dialysis centers. The project is funded by the Patient Centered Outcomes Research Institute (PCORI), a non-profit organization chartered by Congress to fund projects to promote patient-centered care.

DETAILED DESCRIPTION:
OBJECTIVES Primary Objective: The HIGHWay project trains dialysis center teams to conduct ACP conversations with patients with kidney failure. Emphasis is on training and supporting the dialysis center social worker to be the team leader for ACP, in collaboration with the nephrologist and other clinicians.

Aims:

1. Implement the HIGHway intervention with a project team consisting of a social worker, nephrologist and nurse at 50 clinics, and train them to conduct ACP using best practices.
2. Assist social workers/nurses to implement ACP into their regular workflow with personal coaching, webinars and multimedia teaching materials.
3. Use a dedicated web-based application software to guide social workers/nurses on the ACP process of patients in dialysis centers and provide resources for holding ACP conversations.
4. Provide ongoing coaching through monthly teleconferences to bolster social worker/nurse skills through case discussion and mentoring.
5. Develop a long-term implementation and scale-up plan for training social workers/nurses in ACP in different dialysis centers in conjunction with the Coalition for Supportive Care of Kidney Patients, Forum of ESRD Networks, the National Council of Nephrology Social Workers, the National Renal Administrators Association, and dialysis organizations.

RELEVANT BACKGROUND Patient-centered care problem addressed: Patients on dialysis want to discuss their preferences for treatment at the end of life, but few do so, and most nephrologists are reluctant or feel unprepared to lead such discussions. Effective tools are critically needed to elicit such preferences since over 50,000 Americans die of kidney disease annually, more than from breast or prostate cancer. For dialysis patients with significant co-morbidities, risk of death within a year of starting dialysis is stark. Of those who had 4 or more comorbidities, 26% died within 30 days of dialysis initiation, and 60% died within a year. These patients have higher - and often unwanted - intensity of care at end of life; in a four-year study of the United States Renal Data System, 49% of elderly long-term hemodialysis (HD) patients spent time in an intensive care unit in their final month of life, compared with 24% of cancer patients. Meaningful end-of-life conversations can change these outcomes and are associated with increased hospice referral, less aggressive and expensive medical treatment, and higher levels of family satisfaction. Yet less than 10% of end-stage renal disease (ESRD) patients report having a conversation about any end-of-life issues with their nephrologist in the previous year, although 90% said such conversations were important. Few patients with ESRD engage in ACP, and the vast majority lack a written advance directive or surrogate decision maker, leaving them unprepared to provide guidance in medical decisions in a crisis.

A prior study funded by PCORI developed and tested an intervention to enable more advance care planning to take place in dialysis centers. The Shared Decision Making - Renal Supportive Care (SDM-RSC) study tested a multi-modal patient-centered intervention to improve advance care planning for dialysis patients. Through qualitative interviews with advisory boards comprised of patients and stakeholders, SDM-RSC investigators designed an intervention that focused on goals of care conversations between patients and family members with the nephrologist and social worker. The SDM-RSC intervention targeted deficiencies in communication, estimating prognosis, and transition planning for seriously ill dialysis patients. The intervention showed capacity to increase substantially completion of advance directives and medical orders (Medical Orders for Life-Sustaining Treatment [MOLST]/Physician Orders for Life-Sustaining Treatment [POLST]) associated with improved patient-level end-of-life (EOL) outcomes. Among study participants, the advance directive completion rate and understanding of advance directives were substantially higher than in usual care; 75% of participants named and documented a healthcare proxy and 63% had medical orders (MOLST or POLST) (in comparison to 49% with advance directives and 3% with medical orders in usual care). The average duration time for an ACP conversation was about 45 minutes. Overall clinic-level hospice usage using retrospective data did not vary significantly between the pre- and post-intervention 6-month periods with an observed average rate of 25% which is close to the 2015 national average of 26% among all ESRD Medicare decedents. However, among deceased study participants who engaged in a Shared Decision Making and Renal Supportive Care (SDMRSC) meeting, 48% voluntarily withdrew from dialysis prior to death and 39% received hospice services (compared to the overall rate in these dialysis centers of 24.8%).

There were high levels of family satisfaction (FAMCARE results) and no adverse intervention effects on patients or surrogates on measures of depression and health-related quality of life. The stakeholder advisory council and the respondents on post-intervention interviews recommended the following: a) streamlining and focusing the social worker training; b) offering the advance care planning conversation to all dialysis patients, not just those who were seriously ill, c) broadening the population to include home dialysis patients; and d) offering a telehealth option for conducting the discussions.

The current study builds on the SDM-RSC results to implement the revised intervention in a broader population with a larger number of participating dialysis centers.

ELIGIBILITY:
Inclusion Criteria:

* Social worker or nurse must work at a participating dialysis center.
* Social worker, nurse and patients must speak, read and write English.
* All participants must be 18 y old.
* Social workers and nurses Commitment to attend initial 6-h training and booster sessions.

Exclusion Criteria:

* Under 18 years old
* Unable to speak, read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are three separate study populations for this study, with procedures and instruments specific to the population Population 1: Social workers/nurses and dialysis centers will be selected based on demographic data of the center (urbanicity, population served, size of center, patients treated, etc) to provide for diversity of centers participating.
  Population 2: Patients receiving care at the dialysis center where participating social worker/nurses works.
  2a. When an advance care planning conversation takes place, social worker/nurse will provide patient with an informational flyer about the HIGHway project and a postcard.
  2b. Social worker/nurse will identify one patient willing to have a recording made of advance care planning conversation between social worker/nurse and patient.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Advance care conversations attempted, held, documented | During the implementation of the project, one report, year 1
  Patient/Provider Outcome: Self-report of number of conversations social worker has with dialysis patients Self -report of number of conversations social worker has with dialysis patients.
Fidelity of ACP conversations per the HIGHway process taught in trainings | Through implementation completion, one in year 1
  Each social worker will record one ACP conversation with a patient and be assessed on their fidelity to the ACP conversation checklist
Relevance and Significance of ACP intervention for patients | Through implementation completion, one in year 1
  Survey given to patients after an ACP conversation to assess relevance and significance of the conversation to their care

SECONDARY OUTCOMES:
Implementation Outcome: Appropriateness | After finish implementation, one time, year 1
  The perceived fit, relevance, or compatibility of the innovation for a given practice setting, provider, or consumer; to address an issue
Implementation Outcome: Acceptability | Immediately after finish implementation, one in year 1
  Perception that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory.
Characteristics of HIGHway Approach | Immediately after finish implementation, one in year 1
  Perceived usefulness of each element of HIGHway
Feasibility of HIGHway | Immediately after finish implementation, one in year 1
  The extent to which HIGHway was successfully used or carried out

CONTACTS AND LOCATIONS:
Overall Officials: Dale Lupu, PhD, Principal Investigator — George Washington University
Locations (3):
- United States (3):
  - DaVita World Headquarters, Denver, Colorado
  - American Renal Associates LLC Corporate Office, Beverly, Massachusetts
  - Fresenius Medical Care Corporate Headquarters, Waltham, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez de Sosa GM, Thamer M, Anderson E, Unruh ML, Lupu DE. Patient-Centered Advance Care Planning in Dialysis: The HIGHWay (Honor Individual Goals and Hopes Way) Initiative. Kidney360. 2025 Apr 25;6(6):957-967. doi: 10.34067/KID.0000000767. PMID 40279178
- [Derived] Rodriguez de Sosa G, Nicklas A, Thamer M, Anderson E, Reddy N, Stevelos J, Germain MJ, Unruh ML, Lupu DE. Implementing Advance Care Planning for dialysis patients: HIGHway project. BMC Palliat Care. 2022 Jul 16;21(1):129. doi: 10.1186/s12904-022-01011-5. PMID 35841019
- See also: PCORI Website Project Page — https://www.pcori.org/research-results/2021/implementing-advance-care-planning-dialysis-patients